CLINICAL TRIAL: NCT06729307
Title: Ondansetron Combined with Dyclonine Hydrochloride to Improve Patient Experience in Unsedated Esophagogastro-duodenoscopy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-OUEGD
Record Dates: First submitted 2024-11-20; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Esophagogastroduodensocopy (EGD) Procedure
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral ondansetron and dyclonine hydrochloride mucilage (Experimental)
  Interventions: Drug: Oral ondansetron and dyclonine hydrochloride mucilage
- dyclonine hydrochloride mucilage only (Other): Patients are treated with only topical pharyngeal anesthesia (dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to endoscopic process), with no antiemetic drug or placebo.
  Interventions: Drug: Dyclonine hydrochloride mucilage

INTERVENTIONS:
Drug: Oral ondansetron and dyclonine hydrochloride mucilage — Patients will take 8 mg oral ondansetron 2 hours prior to EGD process in addition to dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to EGD process.
  Arms: oral ondansetron and dyclonine hydrochloride mucilage
Drug: Dyclonine hydrochloride mucilage — Patients will be instructed to gurgle 10 mL of dyclonine chloride mucilage (0.01 g/mL) and gurgle for 1 minute 15 minutes prior to endoscopic process.
  Arms: dyclonine hydrochloride mucilage only

SUMMARY:
The goal of this clinical trial is to learn if administering ondansetron prior to esophagogastroduodenoscopy (EGD) can alleviate the gagging reflex, nausea and vomiting in Chinese patients undergoing unsedated diagnostic EGD. The main questions it aims to answer are:

Does taking ondansetron prior to EGD reduce the discomfort of patients during the endoscopic process? Does taking ondansetron prior to EGD reduce the intensity of patient gagging and nausea, and the incidence of vomiting ? Researchers will compare premedication of oral ondasetron and topical pharyngeal anesthesia (dyclonine hydrochloride mucilage) with topical pharyngeal anesthesia only to see if ondansetron can exert the above-mentioned effects.

Participants will be treated with one of the following regimens according to the randomization result:

* Oral ondansetron of 8 mg 2 hours prior to endoscopic process and dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to endoscopic process;
* dyclonine hydrochloride mucilage to be gurgled 15 minutes prior to endoscopic process.

After the endoscopic process is finished, patients will be asked to fill in a questionnaire that contains the following items, all measured by NRS 0-10:

* Overall discomfort;
* Intensity of gagging;
* Willingness to undergo unsedated EGD again if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for diagnostic EGD: patients with symptoms in which EGD may influence di-agnosis and/or disease management, including dysphagia, odynophagia, esophageal refluc symptoms, persistent vomiting, gastrointestinal bleeding, and other upper gastrointestinal symptoms.
* Signing a written informed consent.

Exclusion Criteria:

* Contraindications for esophagogastroduodenoscopy.
* History of upper gastrointestinal tract surgery.
* Severe diseases of the heart, kidney, respiratory system, central nervous system, and hematopoietic system.
* Pregnancy.
* Neuropsychiatric disorders, severe depression and severe anxiety.
* Allergy to ondansetron or dyclonine hydrochloride.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Overall discomfort of patients | from the start of the endoscopic process to the end of the endoscopic process
  measured by NRS 0-10 (0 no discomfort, 10 as uncomfortable as can be), in a questionnaire given to patients after the endoscopic process is finished

SECONDARY OUTCOMES:
Intensity of gagging evaluated by patients | from the start of the endoscopic process to the end of the endoscopic process
  measured by NRS 0-10 (0 none, 10 extremely strong), in a questionnaire given to patients after the endoscopic process is finished
Intensity of patient gagging evaluated by endoscopist | from the start of the endoscopic process to the end of the endoscopic process
  measured by NRS 0-10, (0 none, 10 extremely strong) in a questionnaire given to endoscopists after the endoscopic process is finished
Patient willingness to undergo unsedated EGD again | at the end of the endoscopic process
  the willingness of patients to undergo unsedated EGD in the same method again, assessed by NRS 0-10 (0, not willing at all; 10 completely willing).
Endoscopist satisfaction | from the start to the end of the endoscopic process
  satisfaction of endoscopist in this process, assessed by NRS 0-10 (0, not satisfied at all; 10 very satisfied).

IPD SHARING:
Plan to Share IPD: No